CLINICAL TRIAL: NCT05358132
Title: ARM-ED: Advanced Respiratory Monitoring Events in Drug Toxicity - An Emergency Department Feasibility Study of the Utilisation of a Wearable Device in Patients With Sedative Effects of Drugs
Brief Title: ARM-ED: Advanced Respiratory Monitoring Events in Drug Toxicity
Acronym: ARM-ED
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Pneumowave Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: INGN21RM077
Record Dates: First submitted 2022-03-30; First posted 2022-05-03 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Insufficiency; Overdose of Opiate; Sedative Overdose; Sedative Toxicity
MeSH Terms: conditions — Respiratory Insufficiency; Opiate Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- ARM-ED group 1 - Acute toxicity group: Patients attending the Emergency Department with acute sedating drug toxicity
  Interventions: Device: Pneumowave Device placement and data capture
- ARM-ED group 2 - PSA group: Patients undergoing procedural sedation and analgaesia in the Emergency Department
  Interventions: Device: Pneumowave Device placement and data capture

INTERVENTIONS:
Device: Pneumowave Device placement and data capture — Participants in the acute toxicity group will be studied for a period of time during their Emergency Department attendance or in the case of PSA for the duration of their sedation and recovery period.
  Usual care will be provided to the patient with additional period with Pneumowave biosensor placed onto chest and data capture for a period of time whilst patient is in the Emergency Department,

SUMMARY:
There is a drug-related death crisis in Scotland. The majority of these deaths have involved the misuse of opiates (e.g. heroin) and benzodiazepines (e.g. valium) which cause an individual to stop breathing. The Advanced Respiratory Monitoring Events in Drug Toxicity (ARM-ED) study is a study investigating whether a wearable sensor can help detect problems with breathing in patients who have had drugs or medications that may cause this effect. The study will span a year and will study two groups of patients - those who attend with actual or expected respiratory depression secondary to acute drug toxicity and individuals who have undergone procedural sedation and analgaesia in the Emergency Department.

DETAILED DESCRIPTION:
This study aims to assess if it is feasible to collect respiratory waveform data using an advanced respiratory monitoring device named Pneumowave and whether the device is user friendly in terms of nurse, clinician, and patient.

This is an observational cohort study which utilises passive non-invasive data collection. The device, Pneumowave, will be studied in two distinct groups of patients: those who attend with actual or expected respiratory depression secondary to acute drug toxicity (Group 1) and individuals who have undergone procedural sedation and analgaesia (PSA) in the ED (Group 2). Participants will be studied for the duration of their ED attendance or in the case of PSA for the duration of their sedation and recovery period. They will be followed up via electronic notes 28 days later to identify adverse outcome and to link cases to available toxicology screens performed.

The target number of participants in this study is 100. 50 patients who fit group 1 characteristics and 50 patients who fit group 2 characteristics.

Data from Pneumowave will be analysed in parallel with de-identified clinical and vital sign observational data to inform artificial intelligence driven predictive modelling algorithms.

This study will inform on the utilisation and usability of a wearable device for monitoring an individual's respiratory patterns following the effects of sedative drug use. It will add understanding to potential use of such a device to predict the respiratory compromise in the wearer and alert appropriate stakeholders for timely intervention and ultimately prevention of the wearer's morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

Group 1 - Acute toxicity group

* Presentation to ED due to presumed overdose of drug with potential for respiratory depression (intentional, accidental, recreational, therapeutic excess)
* At least one of GCS <15 or respiratory depression or risk of deterioration of GCS or respiration.
* Age >16 years
* Are willing and able to give informed consent or have available next of Kin to provide informed consent on the participant's behalf
* Able (in the Investigators opinion) and willing to comply with all study requirements

Group 2 - PSA group

* Patient undergoing procedural sedation and anaesthesia in ED
* Age >16 years
* Are willing and able to give informed consent
* Able (in the Investigators opinion) and willing to comply with all study requirements
* Can speak and read English

Exclusion Criteria:

Group 1 - Acute toxicity group

* Unable to provide consent and no next of kin to provide consent on participant's behalf
* Impaired consciousness / respiratory suppression most likely due to cause other than acute drug use
* Condition primarily related to alcohol use and no evidence of acute drug use
* Condition due to withdrawal of drugs / alcohol.
* Treating clinician deems patient inappropriate to be included in study

Group 2 - PSA group

* Unable to provide consent
* Treating clinician deems patient inappropriate to be included in study

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The target number of participants in this study is 100. 50 patients who fit group 1 characteristics and 50 patients who fit group 2 characteristics. All patients who fit the below criteria will be potential candidates for the study. They study team will confirm their eligibility and then they will be included.
  Group 1 - Acute toxicity group screening: any patient presenting to the Queen Elizabeth University Hospital (QEUH) ED with overdose of sedating drug.
  Group 2 - PSA group screening: and patient undergoing PSA in at QEUH ED
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Length of time device in situ on patient | 1 year
  Absolute length of time device in situ on patient and as proportion of intended length of time of device data capture.
Number of times device removed by patient / other | 1 year
  Number of times device removed total during each study episode.
Proportion of waveform data collected while in situ | 1 year
  Length in time of waveform data collection as proportion of intended length of time of device data capture.

SECONDARY OUTCOMES:
Observation of waveform data from Pneumowave device | Duration of study period, up to 15 months
  Observation of waveform data from Pneumowave device and compare to:
  * Normal care vital signs
  * Continuous monitoring vital signs extracted from patient monitors
Compare Pneumowave respiratory wave patterns to clinical events | Duration of study period, up to 15 months
  Compare Pneumowave respiratory wave patterns to clinical events:
  * Normal respiratory patterns
  * Clinical deterioration
  * Interventions in ED
Compare respiratory waveform patterns and motion artefact data | Duration of study period, up to 15 months
  Compare respiratory waveform patterns and motion artefact data to:
  * GCS
  * Richmond Agitation-Sedation Scale (RASS)

CONTACTS AND LOCATIONS:
Overall Officials: David J Lowe, MBChB BMSc FRCEM, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Emergency Department, Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] EMCDDA. Drug-related deaths and mortality in Europe. Update from EMCDDA expert network July 2019. Available from https://www.emcdda.europa.eu, accessed 09/02/2020
- [Background] National records of Scotland, National Statistics. Drug-related deaths in Scotland in 2019, published 15/12/2020. Available from https://www.nrscotland.gov.uk/, accessed 09/02/2020.
- [Background] Holland KM, Jones C, Vivolo-Kantor AM, Idaikkadar N, Zwald M, Hoots B, Yard E, D'Inverno A, Swedo E, Chen MS, Petrosky E, Board A, Martinez P, Stone DM, Law R, Coletta MA, Adjemian J, Thomas C, Puddy RW, Peacock G, Dowling NF, Houry D. Trends in US Emergency Department Visits for Mental Health, Overdose, and Violence Outcomes Before and During the COVID-19 Pandemic. JAMA Psychiatry. 2021 Apr 1;78(4):372-379. doi: 10.1001/jamapsychiatry.2020.4402. PMID 33533876
- [Background] United Nations Office of Drugs and Crime. World Drug Report 2020 Booklet 1. Available from https://wdr.unodc.org/, Accessed 10/02/2021.
- [Background] World Health Organisation. Opioid overdose. August 2020. Available from: https://www.who.int/, Accessed 10/02/2021
- [Background] Scottish Government. Evidence=-Based Strategies for Preventing Drug-Related Deaths in Scotland, Our Emergency Response. January 2020. Available from https://www.gov.scot/. Accessed 10/02/2021
- [Background] McDonald R, Strang J. Are take-home naloxone programmes effective? Systematic review utilizing application of the Bradford Hill criteria. Addiction. 2016 Jul;111(7):1177-87. doi: 10.1111/add.13326. Epub 2016 Mar 30. PMID 27028542
- [Background] Giglio RE, Li G, DiMaggio CJ. Effectiveness of bystander naloxone administration and overdose education programs: a meta-analysis. Inj Epidemiol. 2015 Dec;2(1):10. doi: 10.1186/s40621-015-0041-8. Epub 2015 May 22. PMID 27747742
- [Background] Leino K, Mildh L, Lertola K, Seppala T, Kirvela O. Time course of changes in breathing pattern in morphine- and oxycodone-induced respiratory depression. Anaesthesia. 1999 Sep;54(9):835-40. doi: 10.1046/j.1365-2044.1999.00946.x. PMID 10460553
- [Background] Chu M, Nguyen T, Pandey V, Zhou Y, Pham HN, Bar-Yoseph R, Radom-Aizik S, Jain R, Cooper DM, Khine M. Respiration rate and volume measurements using wearable strain sensors. NPJ Digit Med. 2019 Feb 13;2:8. doi: 10.1038/s41746-019-0083-3. eCollection 2019. PMID 31304358
- [Background] Winhusen T, Theobald J, Lewis D, Wilder CM, Lyons MS. Development and initial testing of a tailored telephone intervention delivered by peers to prevent recurring opioid-overdoses (TTIP-PRO). Health Educ Res. 2016 Apr;31(2):146-60. doi: 10.1093/her/cyw010. PMID 27004905
- [Background] Nandakumar R, Gollakota S, Sunshine JE. Opioid overdose detection using smartphones. Sci Transl Med. 2019 Jan 9;11(474):eaau8914. doi: 10.1126/scitranslmed.aau8914. PMID 30626717
- [Background] Medical research Council , Biomedical Catalyst. 2021. Available from: https://mrc.ukri.org/funding/science-areas/translation/biomedical-catalyst/
- [Background] McDonald R, Campbell ND, Strang J. Twenty years of take-home naloxone for the prevention of overdose deaths from heroin and other opioids-Conception and maturation. Drug Alcohol Depend. 2017 Sep 1;178:176-187. doi: 10.1016/j.drugalcdep.2017.05.001. Epub 2017 May 25. PMID 28654870
- [Background] Community Management of Opioid Overdose. Geneva: World Health Organization; 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK264311/ PMID 25577941
- [Background] EMCDDA (2018) Preventing overdose deaths in Europe.
- [Background] National Institute for Drug Abuse (2017) Naloxone for Opioid Overdose: Life Saving Science. Available online at: https://www.drugabuse.gov/publications/naloxone-opioid-overdose-life-saving-science/naloxone-opioid-overdose-life-saving-science
- [Background] Bird SM, McAuley A. Scotland's National Naloxone Programme. Lancet. 2019 Jan 26;393(10169):316-318. doi: 10.1016/S0140-6736(18)33065-4. No abstract available. PMID 30696566